CLINICAL TRIAL: NCT03857685
Title: Bilateral and Age-dependent Differences in Posterior Capsule Opacification in Vivo Compared to an In-vitro Mode
Brief Title: LEC Proliferation in Vivo and In-vitro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: Proliferation
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Posterior Capsule Opacification
Keywords: Lens capsule; Proliferation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proliferation in an in-vitro model: An in-vitro model is used to study lens epithelial cell proliferation
  Interventions: Procedure: In-vitro model

INTERVENTIONS:
Procedure: In-vitro model — In-vitro model of posterior capsule opacification by culturing the lens capsule

SUMMARY:
Investigate the proliferative capacity of individual lens epithelium capsule specimens in vitro and correlate it to the risk of developing PCO

DETAILED DESCRIPTION:
Cataract, the clouding of the eye's lens, is still the leading cause of blindness worldwide. Until now surgery is the only therapy available for the disease. Cataract surgery is nowadays considered a safe and efficient therapy. However, one of the most frequent complications of cataract surgery is posterior capsule opacification (PCO), which results in diminished postoperative visual acuity. PCO occurs due to a robust wound-healing response, where remaining lens epithelial cells in the capsular bag start to migrate and proliferate.

The lens capsule is divided into an anterior, an equatorial, and a posterior region. The anterior and the equatorial region consist of a single layer of cuboidal epithelial cells, whilst the posterior region is formed of fibers. In the adult lens proliferation occurs almost exclusively in the equatorial region and although the central part of the lens epithelium exhibits very low mitotic activity, it was shown in experiments that cell in this area are also stem cells. There are three possible reasons for the generation of PCO: intraoperative factors (dependening on the amount of remaining cells in the capsular bag), intraocular lens factors, and interpersonal factor (patient-specific factors).

Aim of this study is the generation of an in-vitro model of posterior capsule opacification. Therefore, the investigators will analyse the proliferative capacity of lens epithelial cells on the lens capsule, which is removed during cataract surgery, in a cell culture model. The investigators then compare the proliferative capacity between young and old patients, between both eyes of the same patient, and in different forms of cataract.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract.
* Patients in the age group of 21 years and older.
* Patients with uncomplicated cataract.
* Patients without any relevant systemic or ocular morbidity.
* Patients with well dilating pupils.
* Written informed consent prior to any study specific action.

Exclusion Criteria:

* Patients with complicated cataract.
* Patients with big differences in LOCS scale between the two eyes.
* Patients having corneal pathology.
* Patients with any form of ocular inflammation.
* Patients with glaucoma, retinal pathologies.
* Patients with traumatic cataracts, subluxated and dislocated lens, prior h/o ocular surgery, pseudoexfoliation.
* Any intraoperative complications like posterior capsule rupture.
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age).

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cataract surgery
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Amount of proliferation of lens epithelial cells (LECs) in-vitro compared to in vivo in the same patient | 24 months
  Proliferation of LECs in-vitro will be measured as area/mm2 and correlated with ratings of posterior capsular opacification in vivo using a scale from 0 to 10

SECONDARY OUTCOMES:
Amount of proliferation of LECs in-vitro in young and older patients | 24 months
  Proliferation of LECs in-vitro will be measured as area/mm2 and compared between older and younger individuals
Amount of proliferation of LECs in-vitro between different forms of cataract | 24 months
  Proliferation of LECs in-vitro will be measured as area/mm2 and compared between the different forms of cataract (cortical, nuclear, posterior subcapsular)

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided